CLINICAL TRIAL: NCT02605655
Title: Phase 0 Clinical Trial of Chinese Formula AMP-1915 on Metabolic Syndrome
Brief Title: Clinical Trial of Chinese Formula AMP-1915 on Metabolic Syndrome
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ShanghaiUTCM-01
Record Dates: First submitted 2015-10-22; First posted 2015-11-16 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2014-11

CONDITIONS: Metabolic Syndrome X
Keywords: obesity; hyperlipidemia; hyperglycemia
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Hyperlipidemias; Hyperglycemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMP-1915 (Experimental): Instant noodles contained AMP-1915 2 g/pc with meal, 1 pc/day for 3 months.
  Interventions: Drug: AMP-1915
- Placebo (Placebo Comparator): Instant noodles with the same sharp and color as Experimental noodles with meal, 1 pc/day for 3 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AMP-1915 — A traditional Chinese Formula extract from Astragalus, Radix Puerariae and Cortex Mori is mixed into instant noodles. Patients are treated with AMP-1915 as meal.
  Other Names: Huangqi San
  Arms: AMP-1915
Other: Placebo — Instant noodles without drug
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether the Chinese formula AMP-1915 has effect on Metabolic Syndrome (MS) in MS patients. Half of patients received AMP-1915, while the other half received placebo.

DETAILED DESCRIPTION:
In China, the herbal formulas have been used in the treatment of diabetes for centuries. Huangqisan, investigators named it AMP-1915, is one of traditional Chinese herbal formula used to relieve diabetes which was recorded in Shengji Zonglu (General Medical Collection of Royal Benevolence) published in 1117 A.D. AMP-1915 consists of three herbs: Radix Astragali (roots of Astragalus membranaceus (Fisch.) Bge. var. mongholicus (Bge.) Hsiao, A), Mori Cortex radices (root barks of Morus alba L., M) and Puerariae Lobatae Radix (roots of Pueraria lobata (Willd.) Ohwi., P). Recent studies have shown that these three herbs and their constituents have therapeutic effects on the metabolic disorders.

This randomized, double-blind, placebo-controlled trial was conducted in a community hospital of Shanghai, China. 60 adult participants were metabolic disorder patients according with at least two impaired metabolic profiles (obesity, hyperglycemia, hyperlipidemia or others). During 3-month treatment, participants were randomly divided in to two groups assigned to take AMP-1915 or placebo. AMP-1915 or placebo was mixed into instant noodles as daily meals with same color, shape, size and packaging. BMI, fasting blood glucose (FBG), triglyceride (TG), total cholesterol (TCH), high-density lipoprotein cholesterol (HDL-c), low-density lipoprotein cholesterol (LDL-c), insulin, HbA1c were measured before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Overweight (BMI >= 20) or
* Hyperglycemia (FBG>=6.7 mmol/l) or
* Hyperlipidemia (TG >=1.7 mmol/l or TCH>=5.72 mmol/l or HDL-c <=1.00 mmol/l or LDL-c>=3.12 mmol/l)

Exclusion Criteria:

-

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Fasting blood glucose (FBG) | Change from baseline FBG at 3 months
  Patients' FBG from both placebo and AMP-1915-treated group was collected before treatment as a baseline and after 3-month treatment.
  The difference between these two time points presents the drug effect.

SECONDARY OUTCOMES:
Plasma lipid levels | Change from baseline lipid levels at 3 months
  Patients' blood from both placebo and AMP-1915-treated group was collected before treatment as a baseline and after 3-month treatment. Triglyceride (TG), total cholesterol (TCH), high-density lipoprotein cholesterol (HDL-c), low-density lipoprotein cholesterol (LDL-c) were measured.
  The difference between these two time points presents the drug effect, separately.
Plasma Insulin concentration | Change from baseline insulin concentration at 3 months
  Patients' insulin concentration from both placebo and AMP-1915-treated group was collected before treatment as a baseline and after 3-month treatment.
  The difference between these two time points presents the drug effect.
Body weight | Change from baseline body weight at 3 months
  Patients' body weight from both placebo and AMP-1915-treated group was measured before treatment as a baseline and after 3-month treatment.
  The difference between these two time points presents the drug effect.
Plasma HbA1c | Change from baseline Plasma HbA1c at 3 months
  Patients' Plasma HbA1c from both placebo and AMP-1915-treated group was measured before treatment as a baseline and after 3-month treatment.
  The difference between these two time points presents the drug effect.

CONTACTS AND LOCATIONS:
Overall Officials: Guang Ji, MD, Principal Investigator — Shanghai University of TCM